CLINICAL TRIAL: NCT06058364
Title: A Randomized, Double Blind, Placebo Controlled Parallel Study to Assess the Effects of a Triglyceride on Adults with Low to Moderately Low Mood.
Brief Title: Effect of a Nutritional Supplement on Mental Wellness in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmavite LLC (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AFCRO-163
Record Dates: First submitted 2023-09-08; First posted 2023-09-28 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Low Mood
Keywords: triglyceride; fatty acids; mental wellness; mood; microbiome; gut-brain axis; dietary supplement
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: This is a double-blind randomized placebo controlled trial for a dietary supplement with two parallel groups - triglyceride supplement and placebo.
Who Masked: Participant, Investigator
Masking Description: Blinding of both study team and participants will be ensured by only providing access to the randomization list to the science and quality team. The relationship between the randomization number and the group assignment will be unknown to the participants, clinical study team, and the Sponsor, i.e. the study will be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention 1 (Experimental): Participants receiving triglyceride supplement
  Interventions: Dietary Supplement: Intervention 1 - Triglyceride
- Intervention 2 (Placebo Comparator): Participants receiving placebo
  Interventions: Dietary Supplement: Intervention 2 - Placebo

INTERVENTIONS:
Dietary Supplement: Intervention 1 - Triglyceride — Triglyceride (1 softgel each morning with a glass of water)
  Arms: Intervention 1
Dietary Supplement: Intervention 2 - Placebo — Placebo (1 softgel each morning with a glass of water)
  Arms: Intervention 2

SUMMARY:
Trillions of microbes reside in human gut and constitute "gut microbiota". Composition of these microbes and substances produced by them play an important role in human health and wellness.

The goal of this study is to determine if a unique orally consumed triglyceride supplement will impart mood benefits. Investigators hypothesize that a part of the fatty acids will be released in upper gastrointestinal (GI) tract and can be absorbed and reach different organs via systemic circulation (blood), including to the brain, and provide health benefits. Rest of the portion would reach the colon and may modulate gut microbiota and provide health benefits via the gut-brain axis (a bi-directional communication between emotional and cognitive centers and the gastrointestinal system). These health benefits could include alleviation of stress, occasional anxiousness and low mood.

Participants with self-reported low mood will be randomized to two groups - one group will receive triglyceride supplement in softgel form and another group will receive a placebo (softgel with no active substance). Investigators will evaluate the effect of consumption of triglyceride supplement compared to Placebo on occasional low mood, occasional anxiousness, stress, sleep and general health by measuring changes from baseline.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, parallel study, which will include 5 visits over 10 week period - a screening visit (Visit 1; week -3), a 3-week run-in period followed by baseline determination or baseline visit (Visit 2; day 0), and three test visits (Visits 3, 4, and 5 at days 14, 28, and 56 respectively).

SCREENING

Visit 1 - Week -3

At Visit 1 (Screening visit) Participants will attend the study site and the following procedures will be carried out:

* Participants will receive oral and written information about the study and be allowed to ask questions.
* Participants will sign the informed consent document.
* Inclusion and exclusion criteria will be reviewed.
* Demographic, health, and lifestyle data will be collected.
* Medical history will be collected.
* Concomitant medication will be recorded.
* Height and weight will be measured, and Body Mass Index (BMI) calculated.
* Vitals (blood pressure, heart rate and temperature) will be recorded.
* Complete Block Fiber screener
* Download the Electronic Patient Reported Outcomes (ePRO) questionnaire app to the participants device.
* Complete Hospital Anxiety and Depression (HADS) questionnaire.
* A blood sample will be collected for screening and safety analysis.
* For participants of childbearing potential, a urine sample will be collected, and pregnancy test performed (regardless of contraceptive use or relationship status).
* Participants will be provided with a stool collection kit and instructions for collecting and storing their sample. Participants will collect a stool sample at home, within 48 hours of their scheduled visit and bring it to the clinic at their next visit.
* Participants will be provided with a saliva collection kit and instructions for collecting and storing their sample. Participants will collect a saliva sample at home, at T0, T30, T45, T60 minutes after waking on the morning of their scheduled visit and bring it to the clinic at their visit.
* Participants will be provided with the Karolinska Sleepiness Scale (KSS). Participants will complete this 5 minutes after collecting T0 saliva sample on the morning of their scheduled visit and bring it to the clinic at their visit.
* Participants will be provided with a 3-day food diary and instructions on how to complete the document. Participants will return their completed diary at their next visit.
* Participants will be reminded to complete the questionnaires with 24 hours of their next visit.
* Participants will be provided with a provisional appointment to attend a Dual X-ray absorptiometry (DEXA) scan.

Participants will be given an appointment to return to the study site within 21 days for their baseline/day 1 visit.

INTERVENTION PHASE

Visit 2 - Day 0

Participants will complete a dual X-ray absorptiometry (DEXA) scan in advance of taking their first dose of study product, between Day -21 and Day 0.

Participants will attend this study visit and the following procedures will be carried out:

* Participant's continued consent to study procedures will be confirmed.
* Inclusion/exclusion criteria will be reviewed.
* Adverse events will be recorded.
* Concomitant medication/supplements will be recorded.
* Weight will be measured, and BMI calculated.
* Vitals (blood pressure, heart rate and temperature) will be recorded.
* For individuals of childbearing potential, a urine sample will be collected, and pregnancy test performed (regardless of contraceptive use or relationship status).
* Participants will return their saliva samples and samples will be stored for future analysis.
* Participants will return their stool sample and sample will be stored for future analysis.
* Participants will return their completed 3-day food diary.
* Participants will return their completed Karolinska Sleepiness Scale (KSS) questionnaire.
* Participants will have completed the following questionnaires within 24 hours of the visit:

  * Cohen's Perceived Stress Scale (PSS)
  * 36 item short form survey (SF-36)
* Complete Hospital Anxiety and Depression (HADS) questionnaire.
* A blood sample will be collected and stored for future biomarker analysis.
* Participants will be provided with a stool collection kit and instructions for collecting and storing their sample. Participants will collect a stool sample at home, within 48 hours of their scheduled visit and bring it to the clinic at their next visit.
* Participants will be provided with a saliva collection kit and instructions for collecting and storing their sample. Participants will collect a saliva sample at home, at T0, T30, T45, T60 minutes after waking on the morning of their scheduled visit and bring it to the clinic at their visit.
* Participants will be provided with the Karolinska Sleepiness Scale (KSS). Participants will complete this 5 minutes after collecting T0 saliva sample on the morning of their scheduled visit and bring it to the clinic at their visit.
* Participants will be reminded to complete the questionnaires with 24 hours of their next visit.
* Participants will be provided with a watch for monitoring their sleep and instructions for how to wear and use the watch.

Participants will be randomized into one of two treatment groups as follows, but will be blinded as to which group, they are in:

* Group 1: Triglyceride supplement
* Group 2: Placebo

Participants will be supplied with an 8-week supply of study product and instructions of dosing. Participants will be instructed to take one soft-gel capsule each day for the next eight weeks. An additional eight days of doses will be supplied in case of delay of study visit or loss of study product.

- Participants will be provided with an appointment to return to the study site in two weeks.

Visit 3 - Day 14

Participants will return to the study site at day 14 and the following procedures will be carried out:

* Participant's continued consent to study procedures will be confirmed.
* Adverse events will be recorded.
* Concomitant medication/supplements will be recorded.
* Data from the Participant's sleep watch will be reviewed and battery for the watch will be replaced.
* Participants will return their saliva samples and samples will be stored for future analysis.
* Participants will return their stool sample and sample will be stored for future analysis.
* Participants will return their completed KSS questionnaire.
* Participants will have completed the following questionnaires within 24 hours of the visit:

  * 36 item short form survey (SF-36)
* Complete Hospital Anxiety and Depression, HADS questionnaire.
* A blood sample will be collected and stored for future biomarker analysis.
* Participants will be provided with a stool collection kit and instructions for collecting and storing their sample. Participants will collect a stool sample at home, within 48 hours of their scheduled visit and bring it to the clinic at their next visit.
* Participants will be provided with a saliva collection kit and instructions for collecting and storing their sample. Participants will collect a saliva sample at home, at T0, T30, T45, T60 minutes after waking on the morning of their scheduled visit and bring it to the clinic at their visit.
* Participants will be provided with the Karolinska Sleepiness Scale (KSS). Participants will complete this 5 minutes after collecting T0 saliva sample on the morning of their scheduled visit and bring it to the clinic at their visit.
* Participants will be reminded to complete the questionnaires with 24 hours of their next visit.
* Participants will be provided with an appointment to return to the study site in two weeks.

Visit 4 - Day 28

Participants will return to the study site at day 28 and the following procedures will be carried out:

* Participant's continued consent to study procedures will be confirmed.
* Adverse events will be recorded.
* Concomitant medication/supplements will be recorded.
* Data from the Participant's sleep watch will be reviewed and battery for the watch will be replaced.
* Participants will return their saliva samples and samples will be stored for future analysis.
* Participants will return their stool sample and sample will be stored for future analysis.
* Participants will return their completed Karolinska Sleepiness Scale (KSS) questionnaire.
* Participants will have completed the following questionnaires within 24 hours of the visit:

  * Cohen's Perceived Stress Scale (PSS)
  * 36 item short form survey (SF-36)
* Complete Hospital Anxiety and depression (HADS) questionnaire.
* A blood sample will be collected and stored for future biomarker analysis.
* Participants will be provided with a stool collection kit and instructions for collecting and storing their sample. Participants will collect a stool sample at home, within 48 hours of their scheduled visit and bring it to the clinic at their next visit.
* Participants will be provided with a saliva collection kit and instructions for collecting and storing their sample. Participants will collect a saliva sample at home, at T0, T30, T45, T60 minutes after waking on the morning of their scheduled visit and bring it to the clinic at their visit.
* Participants will be provided with the Karolinska Sleepiness Scale (KSS). Participants will complete this 5 minutes after collecting T0 saliva sample on the morning of their scheduled visit and bring it to the clinic at their visit.
* Participants will be reminded to complete the questionnaires with 24 hours of their next visit.
* Participants will be provided with a 3-day food diary and instructions on how to complete the document. Participants will return their completed diary at their next visit.
* Participants will be provided with an appointment to return to the study site in two weeks.

Visit 5 (Final Visit) - Day 56

Participants will return to the study site at day 56 and the following procedures will be carried out:

* Adverse events will be recorded.
* Concomitant medication/supplements will be recorded.
* Participants will return any unused study product and compliance will be assessed.
* Participants will return their sleep watch and the data from the Participant's sleep watch will be reviewed.
* Participants will return their saliva samples and samples will be stored for future analysis.
* Participants will return their stool sample and sample will be stored for future analysis.
* Participants will return their 3-day food diary.
* Participants will return their completed Karolinska Sleepiness Scale (KSS) questionnaire.
* Weight will be measured, and BMI calculated.
* Vitals (blood pressure, heart rate and temperature) will be recorded.
* Participants will have completed the following questionnaires within 24 hours of the visit:

  * Cohen's Perceived Stress Scale (PSS)
  * 36 item short form survey (SF-36)
* Complete Hospital Anxiety and Depression (HADS) questionnaire.
* The questionnaire data will be reviewed, and the app deleted from the participants device.
* A blood sample will be collected for safety analysis.
* A blood sample will be collected and stored for future biomarker analysis.
* For participants of childbearing potential, a urine sample will be collected, and pregnancy test performed (regardless of contraceptive use or relationship status)
* Participants will attend a DEXA scan 0 to 7 days after Visit 5.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, the Participant must fulfil all the following criteria:

1. Be willing to participate in the study and comply with its procedures.
2. Be able to give written informed consent.
3. Adults aged between 18 and 65 years (inclusive).
4. Participants with a BMI between ≥18.5 and <30.0 kg/m^2.
5. Has self-reported mild-moderate low mood, confirmed by a Hospital Anxiety and Depression Scale (HADS - D) score 8 - 14.
6. Be willing to maintain stable dietary habits and physical activity levels throughout the study period.
7. Be able to communicate well with the Investigator, to understand and comply with the requirements of the study and be judged suitable for the study in the opinion of the Investigator.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. Recent use of probiotics, prebiotics, postbiotic and other fermented foods that contain live bacteria within last 30 days from Visit 2.
2. Recent use of any dietary supplements, within last 14 days from Visit 2.
3. Participant who has been on antibiotics during the 90 days from Visit 2.
4. Participant with a malignant disease or any concomitant end-state organ disease and/or laboratory abnormalities considered by Investigators to be risky or that could interfere with data collection.
5. Participants who have started receiving cognitive behavioural therapy (CBT) or psychotherapy in the last 90 days prior to Visit 2 or plan to start during the period of the study.
6. Participant who is severely immunocompromised (HIV positive, transplant patient, on anti-rejection medications, on a systemic steroid treatment for >30 days, or chemotherapy or radiotherapy within the last year).
7. Significant psychiatric diagnosis (e.g., bipolar), as diagnosed by a healthcare professional, including major depressive disorder (e.g., clinical depression) and anxiety disorder.
8. Participants taking anti-depressants or herbal treatments for mood disorders or psychological conditions (e.g., valerian, St. John's Wort) within 90 days prior to Visit 2 or planning to start during the study period.
9. Participants who are on anxiolytics, antipsychotics, anticonvulsants, antidepressants, opioid pain relievers, hypnotics, and/or prescribed sleep medication within 30 days prior to screening (Visit 1).
10. Participants with a current history of drug (including illicit drug) and /or alcohol abuse at the time of enrolment.
11. Participants who consume any products containing Tetrahydrocannabinol (THC) and Cannabidiol (CBD) 30 days prior to screening (Visit 1).
12. Participants who are unwilling to only consume butter or margarine once per day for the duration of the study.
13. Participants with a fiber intake of >18g/day
14. Participants who are pregnant (determined by urine pregnancy test for all individuals of childbearing potential at screening, regardless of contraceptive use or relationship status), breastfeeding, or wish to become pregnant during the study.
15. Have an acute or chronic illness (e.g., heart disease, uncontrolled hypertension, uncontrolled hypercholesterolemia, inflammatory bowel disease, cancer, HIV) that, in the Investigators judgment, precludes involvement in the study.
16. Have had any other condition or are taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk, or confound the interpretation of the study results.
17. Change in prescribed medication, or major diet change in the 30 days prior to enrolment (Visit 2).
18. Has received treatment involving experimental drugs in the past 90 days and experimental supplements in the past 60 days at the discretion of the investigator.
19. Individuals who, in the opinion of the investigator, are considered to be poor clinical attendees or unlikely for any reason to be able to comply with the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of eight weeks consumption of triglyceride supplement compared to Placebo on low mood in a population with self-reported mild to moderate symptoms (Hospital Anxiety and Depression Scale - Depression, HADS-D score of 8 - 14). | From baseline to Week 8
  A change in self-reported symptoms of low mood assessed by Hospital Anxiety and Depression Scale - Depression (HADS-D) at baseline to week 8. HADS-D sub-score ranges from 0 - 21, where higher score is worse.

SECONDARY OUTCOMES:
To evaluate the effect of consumption of triglyceride supplement compared to Placebo on low mood, in a population with self-reported mild to moderate symptoms (Hospital Anxiety and Depression Scale - Depression (HADS-D) score of 8 - 14). | From baseline to week 2 and week 4
  A change from baseline to week 2 and week 4, in self-reported mild to moderate symptoms assessed by Hospital Anxiety and Depression Scale, HADS Depression sub score (HADS-D), .which ranges from 0 - 21 and higher score is worse.
To evaluate the effect of consumption of triglyceride supplement compared to Placebo in a population with self-reported low mood with mild to moderate symptoms on anxiety. | From baseline to weeks 2, 4 and 8
  A change from baseline to weeks 2, 4 and 8 in self-reported anxiety assessed by Hospital Anxiety and Depression Scale, HADS anxiety sub score (HADS-A).HADS-A sub score range from 0 - 21, where higher score is worse.
To evaluate the effect of consumption of triglyceride supplement compared to Placebo in a population with self-reported low mood with mild to moderate symptoms on sleep using Motionlogger Micro Watch (Sleep Watch) and Karolinska Sleepiness Scale (KSS). | From baseline to weeks 2, 4 and 8
  1. A change from baseline to weeks 2, 4 and 8 in activity index score recorded by Sleep Watch.
  2. A change from baseline to weeks 2, 4 and 8 in total duration in bed (min) recorded by Sleep Watch.
  3. A change from baseline to weeks 2, 4 and 8 in latency to persistent sleep (min) recorded by Sleep Watch.
  4. A change from baseline to weeks 2, 4 and 8 in sleep efficiency (%) recorded by Sleep Watch.
  5. A change from baseline to weeks 2, 4 and 8 in sleep fragmentation (events/h) recorded by Sleep Watch.
  6. A change from baseline to weeks 2, 4 and 8 in sleep minutes (min) recorded by Sleep Watch.
  7. A change from baseline to weeks 2, 4 and 8 in wake after sleep onset (WASO) (min) recorded by Sleep Watch.
  8. A change from baseline to weeks 2, 4 and 8 in perceived awakening refreshed level assessed by Karolinska Sleepiness Scale (KSS) Score for waking up refreshed. KSS is a 9 point scale (1 - 9), where 1 = extremely alert and 9 = extremely sleepy)
To evaluate the effect of consumption of triglyceride supplement compared to Placebo in a population with self-reported low mood with mild to moderate symptoms on general health, physical functioning and energy | From baseline to weeks 2, 4 and 8 or weeks 4 and 8
  Short -Form 36 score ranges from 0 - 100. Higher scores indicate higher quality of life.
  1. A change from baseline to weeks 2, 4 and 8 in quality of life as measured by Short-Form 36 general health scale.
  2. A change from baseline to weeks 2, 4 and 8 in quality of life as measured by Short-Form 36 physical functioning scale.
  3. A change from baseline to 4 and 8 in quality of life as measured by Short-Form 36 energy/fatigue scale.
To evaluate the effect of consumption of triglyceride supplement compared to Placebo in a population with self-reported low mood with mild to moderate symptoms on Stress | From baseline to weeks 4 and 8
  A change from baseline to weeks 4 and 8 in perceived stress level assessed by Cohen's Perceived Stress Scale (PSS). Cohen's Perceived Stress Scale ranges from 0 - 40. Higher scores indicate greater perceived stress levels.
To evaluate the effect of consumption of triglyceride supplement compared to Placebo in a population with self-reported low mood with mild to moderate symptoms on salivary cortisol | From baseline to weeks 2, 4 and 8
  1. A change from baseline to weeks 2, 4 and 8 in salivary cortisol (nmol/L) from T0 to post awakening samples T30
  2. A change from baseline to weeks 2, 4 and 8 in salivary cortisol (nmol/L) from T0 to post awakening samples T45
  3. A change from baseline to weeks 2, 4 and 8 in salivary cortisol (nmol/L) from T0 to post awakening samples T60
  4. A change from baseline to weeks 2, 4 and 8 in salivary cortisol (nmol/L) awakening response (CAR) as measured by Area Under the Curve (AUC) (T0, T30, T45, T60).

OTHER OUTCOMES:
To evaluate the effect of consumption of triglyceride supplement compared to Placebo in a population with self-reported low mood with mild to moderate symptoms on fat mass measured by dual X-ray absorptiometry (DEXA) | From baseline to 8 weeks
  A change from baseline to week 8 in fat mass as a percentage of total mass (%).
To evaluate the effect of consumption of triglyceride supplement compared to Placebo in a population with self-reported low mood with mild to moderate symptoms on gut microbial composition | From baseline to 8 weeks
  A change from baseline to week 8 in gut microbial composition as determined by shot gun sequencing of fecal DNA

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Clinical Trials, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No